CLINICAL TRIAL: NCT01707537
Title: Phase I Study to Determine the Safety and Immunogenicity of Euvichol(Oral Cholera Prevention Vaccine)in Healthy Adult Men ; Open, Non-comparative Clinical Trial
Brief Title: To Determine the Safety and Immunogenicity of an Oral(Whole Cell) Euvichol Cholera Vaccine in Healthy Adult Men
Acronym: OCV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Collaborators: Instituto Universitario IVI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UBC101
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Prevention Harmful Effects
Keywords: OCV; cholera
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Euvichol (Experimental): Euvichol is a homogeneous suspension of inactivated suitable strains of Vibrio cholera serogroup O1 and O139. Euvichol is Yellow to yellowish colour.
  Interventions: Biological: Euvichol

INTERVENTIONS:
Biological: Euvichol — 1.5mL/vial, 1vial at 2-week intervals twice
  Other Names: Oral Cholerae Vaccine

SUMMARY:
To Determine the Safety and Immunogenicity of an Oral(Whole Cell) Euvichol Cholera Vaccine in Healthy Adult Men

DETAILED DESCRIPTION:
This clinical trial is open, non-comparative phase 1 clinical studies in healthy men and has been designed to determine the safety and immunogenicity of Euvichol(Oral cholera vaccine)

ELIGIBILITY:
Inclusion Criteria:

* Adult men over 20years of age
* More than 45kg body weight and ideal body weight within ±20% of the weight
* Screening was conducted within 14 days of investigational drug administration (Vital Sign & Physical Examination, hematology and blood coagulation tests, blood chemistry tests, urinalysis, 12-lead ECG, etc.), the results at the discretion of the investigator deemed suitable for participation in clinical trials
* Written consent person who determines to participate in a clinical trial

Exclusion Criteria:

* A person who showed hypersensitivity when other preventive vaccination in the past
* A person who have received cholera vaccine in the past
* A person who had a febrile illness or infection disease, or have received antibiotics within 2weeks before the start of the experiment
* A person who had gastrointestinal symptoms such as diarrhea, abdominal pain, or have been received prescription drug within one week before the start of the experiment
* A person who was lasted for more than two weeks of symptoms such as diarrhea, abdominal pain within 6months before the start of the experiment
* A person who donate whole blood or component of blood within one months before the start of the experiment if the donors
* A person who received other preventive vaccine within 2months before the start of the experiment
* A person who received blood products of immune globulin preparations within 3months before the start of the experiment
* A person who has immune function disorders or are receiving immunosuppressive treatment
* A person who has chronic illness in progress
* Ongoing drug and alcohol abuse(Not more than 28 units/week for drinking)
* A person who participate in clinical trials treated with the investigational drug within 2months before the start of the experiment
* A person who is difficult to participate in this clinical trials as the discretion of the investigator

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety(proportion of subjects with adverse events) | From the date of the first orally administered for 4 weeks after the second dose
  The proportion of all adverse event and serious adverse event which were occured during the entire study period is analyzed and casuality between severity and investigational product is presented.
  Check the vital signs, physical examination and clinical laboratory tests

SECONDARY OUTCOMES:
Immunogenicity(vibriocidal antibody assay) | Baseline(before the administration), 14 days after first dose, 14 days after second dose
  Proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies, relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hong J Hee, Ph.D, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, Chungcheongnam-do, South Korea

REFERENCES:
- [Derived] Baik YO, Choi SK, Kim JW, Yang JS, Kim IY, Kim CW, Hong JH. Safety and immunogenicity assessment of an oral cholera vaccine through phase I clinical trial in Korea. J Korean Med Sci. 2014 Apr;29(4):494-501. doi: 10.3346/jkms.2014.29.4.494. Epub 2014 Apr 1. PMID 24753695